CLINICAL TRIAL: NCT07399730
Title: A Non-interventional Study Evaluating Ravulizumab Treatment Outcomes in Polish Patients With Atypical Hemolytic Uremic Syndrome
Brief Title: Ravulizumab Outcomes in Polish Patients With aHUS
Acronym: aHUS-OPTIMUM
Status: Not yet recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D928BR00003
Record Dates: First submitted 2026-01-27; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Atypical Hemolytic Uremic Syndrome
Keywords: aHUS; Atypical Hemolytic Uremic Syndrome; Ravulizumab; Observational
MeSH Terms: conditions — Atypical Hemolytic Uremic Syndrome | interventions — ravulizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective cohort: Group of patients naive to complement inhibitors
  Interventions: Drug: Ravulizumab
- Retrospective cohort: Group of patients who transitioned from other complement inhibitors to ravulizumab.
  Interventions: Drug: Ravulizumab

INTERVENTIONS:
Drug: Ravulizumab — Ultomiris

SUMMARY:
This multicenter, observational cohort study uses retrospective collection of past medical history and prospective follow-up to capture longitudinal data on the management and clinical outcomes of patients with atypical hemolytic uremic syndrome (aHUS) treated with ravulizumab as part of routine clinical practice under Poland's National Drug Program (NDP).

ELIGIBILITY:
Inclusion Criteria:

* Patients of all ages diagnosed with atypical hemolytic uremic syndrome (aHUS) who received treatment with ravulizumab under the National Drug Program (NDP) in Poland.
* Patients who are willing to participate in the study and have provided informed consent by signing the informed consent form (ICF).

Exclusion Criteria:

* Individuals who intend to participate in a clinical trial for atypical hemolytic uremic syndrome (aHUS) on or after the date of their first ravulizumab infusion through the National Drug Program.
* Patients with cognitive impairments, those who are unwilling to participate, or those facing language barriers that hinder adequate comprehension or cooperation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients naïve to complement inhibitors (prospective cohort) with a body weight of 10 kg or above (no age restrictions) diagnosed with atypical haemolytic uremic syndrome and meeting all ravulizumab treatment eligibility criteria listed in NDP - no previous exposition to CIs including clinical trials, EAP etc.
  Patients who have been switched to ravulizumab from other CI (retrospective cohort) with a body weight of 10 kg or above (no age restrictions) diagnosed with atypical haemolytic uremic syndrome and meeting all ravulizumab treatment eligibility criteria listed in NDP.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patient attaining Complete Thrombotic Microangiopathy (TMA) Response during observation (naïve) | Up to 24 months
  In order to achieve the primary objectives, the following variables will be estimated: To assess ravulizumab primary treatment outcome in Polish patients with aHUS
Proportion of patients attaining/maintaining. Complete TMA Response during observation (switched) | Up to 24 months
  In order to achieve the primary objectives, the following variables will be estimated: To assess ravulizumab primary treatment outcome in Polish patients with aHUS

SECONDARY OUTCOMES:
Time to Complete TMA Response | Up to 24 months
  Time from initiation of ravulizumab to TMA Response: continuous variable (days; specify when complete response criteria are met)
Proportion of dialysis-free patients | Up to 24 months
  In order to achieve the secondary objectives, the following variables will be estimated
Complete TMA response | Up to 24 months
  In order to achieve the secondary objectives, the following variables will be estimated:
  * Platelet count (≥150 x 109/L)
  * Lactate dehydrogenase (LDH) levels (≤ULN)
  * Serum creatinine (≤ULN for age or an improvement > 25% compared to baseline),
Proportion of patients with lab results normalization during observation | Up to 24 months
  Laboratory Parameters:
  * platelet count (≥150 x 109/L)*,
  * lactate dehydrogenase (LDH) levels (≤ULN),
  * serum creatinine (≤ULN for age or an improvement > 25% compared to baseline),
  * serum creatinine improvement of >50% compared to baseline
  * estimated glomerular filtration rate (eGFR) ≥ 60 mL/min/1.73 m2,
  * increase in haemoglobin of ≥ 20 g/L
Change from baseline in CKD stage, as evaluated by the physician over time | Up to 24 months
  In order to achieve the secondary objectives, the following variables will be estimated:
  CKD stage 1 (rather theoretical at baseline, possible following successful treatment): eGFR ≥90 ml/min./1.73m2 CKD stage 2 (rather theoretical at baseline, possible following successful treatment): eGFR 60 - 90 ml/min./1.73m2 CKD stage 3a: eGFR 45 - 59 ml/min./1.73m2 CKD stage 3b: eGFR 30 - 44 ml/min./1.73m2 CKD stage 4: eGFR 15 - 29 ml/min./1.73m2 CKD stage 5: eGFR< 15 ml/min./1.73m2 CKD stage 5D: need for dialysis independent from eGFR value
Change from baseline in proteinuria status over time | Up to 24 months
  In order to achieve the secondary objectives, the following variables will be estimated: At least one of the following numbers describing the highest proteinuria and/or albuminuria:
  * urine protein-to-creatinine ratio [mg/g] (preferred)
  * urine protein loss [mg/24 hours]
  * urine protein concentration [mg/dl]
  * urine albumin-to-creatinine ratio [mg/g] (preferred)
  * urine albumin loss [mg/24 hours]
  Urine protein reduction to ≤ 500 mg/g (500 mg/24 hours) Urine protein reduction by ≥50% from baseline Time to urine protein reduction to ≤ 500 mg/g (500 mg/24 hours) Time to urine protein reduction by ≥50% from baseline
Change from baseline in the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue; adults) and Pediatric Functional Assessment of Chronic Illness Therapy - Fatigue (Peds FACIT-F; pediatric patients) score overtime (naïve) | Up to 24 months
  FACIT-Fatigue - scoring ranges from 0 (highest fatigue) to 52 (lowest fatigue), where higher scores indicate lower levels of fatigue.
  Peds FACIT-F - scoring ranges from 0 (highest fatigue) to 52 (lowest fatigue), where higher scores indicate lower levels of fatigue.
Change form baseline in EQ- 5D-5L (adults) and EQ-5D-Y- 5L (paediatric patients) score overtime (naïve) | Up to 24 months
  EQ-5D-5L/EQ-5D-Y-5L consists of 2 pages: EQ-5D descriptive system and EQ visual analogue scale (EQ VAS).
  EQ-5D/EQ-5D-Y comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems.
  EQ VAS - scale rating from 0 (worst imaginable health state) to 100 (best imaginable health state)

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/